CLINICAL TRIAL: NCT01464281
Title: A Randomized, Multicenter Study Evaluating HBsAg Clearance in CHB Patients Achieving HBeAg Loss and HBV DNA <200copies/ml on Treatment With Nucleotide Analogues and Switched to Peginterferon Alfa-2a
Brief Title: A Study of Switch From Nucleotide to Peginterferon Alfa-2a in CHB Patients Achieving HBeAg Loss and HBV DNA <200IU/ml
Acronym: New Switch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hong Ren, Principal Investigator, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27928
Record Dates: First submitted 2011-10-19; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Hepatitis B
Keywords: nucleoside; peginterferon alfa-2a
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 48-week standard treatment (Experimental): 48-week standard treatment by Peginterferon alfa 2a 180µg/week
  Interventions: Drug: Peginterferon alfa 2a
- 96-week prolonged treatment (Active Comparator): 96-week prolonged treatment by Peginterferon alfa 2a 180µg/week
  Interventions: Drug: Peginterferon alfa 2a

INTERVENTIONS:
Drug: Peginterferon alfa 2a — Group 1 : 48-week standard treatment by Peginterferon alfa 2a 180µg/week Group 2 : 96-week prolonged treatment by Peginterferon alfa 2a 180µg/week.

SUMMARY:
A Randomized, open-label, multicenter study.

The patients after 1-3 years NAs treatment and having achieved HBeAg loss and HBV DNA <200IU/ml will be switched to Pegasys for 48 or 96 weeks (with a 12 weeks period of overlap with the NA for safety reasons). The subjects will be randomized into 2 groups:

Group 1 : 48-week standard treatment by Peginterferon alfa 2a 180µg/week Group 2 : 96-week prolonged treatment by Peginterferon alfa 2a 180µg/week.

All the patients will be followed up for 48 weeks after discontinuation of the study medication.

Note: NAs will be stratified LAM, ETV and ADV, with the ratio 1:1:1.

DETAILED DESCRIPTION:
eligibility criteria: Men and women old of 18 to 65 years with chronic hepatitis B HBeAg positive treated with nucleoside and/or nucleotide analogues for 1-2 years and with partial response (HBeAg loss and HBV DNA <1000copies/ml).

ELIGIBILITY:
Inclusion Criteria:

* Patients on-treatment with NAs (ADV, ETV or LAM) for 1-3 years, having achieved HBeAg loss at screening, and HBV DNA <200IU/ml for at least 48 weeks
* Male and female patients ≥ 18 to 65 years of age
* Chronic hepatitis B (positive HBsAg for at least 6 months prior to NA therapy start)
* Compensated liver disease (Child-Pugh <6)
* Absence of hepatocellular carcinoma on liver imaging and/or alfa fetoprotein < 50 ng/ml
* Negative urine or blood pregnancy test for women of childbearing potential within 24 hours of first PEG IFN study medication administration
* Able and willing to provide informed consent and abide by the requirements of the study

Exclusion Criteria:

* Neutrophil count <1.5 x 109cells/L or platelet count <90 x 109cells/L
* Co-infections with HIV, HAV, HCV, HDV or HEV
* Women with ongoing pregnancy or breast feeding, or wishing to become pregnant during the study period
* Prolonged and excessive alcohol intake (> 40g/day for men and > 30g/day for women)
* Active intravenous drug abuse
* History or current treatment with telbivudine
* Treatment with immunomodulators (e.g. Interferon) for less than one year before study enrollment
* Treatment with immunosuppressors (including systemic corticosteroids) or anti-neoplastic treatment (including radiation therapy) <=6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Serum concentrations of ceruloplasmin or alfa-antitrypsin consistent with an increased risk of metabolic disease
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of severe cardiac disease
* History of the severe seizure disorder or current anticonvulsivant use
* History of thyroid disease poorly controlled on prescribed medications. Patients with elevated thyroid stimulating hormone concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* History or other evidence of severe retinopathy
* History of autoimmune disease or presence of a significant level of auto-antibodies
* Renal insufficiency (creatinine clearance of < 50 ml/min according to the Cockroft and Gault equation), kidney transplant, hemodialysis
* History of depression or uncontrolled psychiatric disorders
* Subjects protected by law or not in a position to give consent
* Patients with reproductive potential not willing to use an effective method of contraception.
* Evidence of an active or suspected cancer or a history of malignancy (other than basocellular carcinoma or in-situ cervical carcinoma)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
determine the response rate (HBsAg clearance at Week 48 and 96) | 1 year
  To determine the response rate (HBsAg clearance at Week 48 and 96) in subjects who are being treated by NAs and achieved a combined response which consists of both HBeAg loss and HBV DNA <1000 copies/ml

SECONDARY OUTCOMES:
HBsAg/HBeAg/HBV DNA changes/ALT normalization /HBsAg seroconversion at EOT and EOF | 1 year
  1. HBsAg loss at EOF
  2. Quantitative HBe/sAg reduction at every check point.
  3. HBeAg seroconversion at EOT and EOF
  4. HBV DNA changes over 48 or 96 weeks at every check points
  5. ALT normalization at EOT and EOF
  6. HBsAg seroconversion at EOT and EOF

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, Principal Investigator — The 2nd affiliated Hospital of Chongqing Medical University
Locations (1):
- The 2nd affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Hu P, Shang J, Zhang WH, Gong GZ, Li YG, Chen XY, Jiang JN, Xie Q, Dou XG, Sun YT, Li YF, Liu YX, Liu GZ, Ma DW, Chi XL, Tang H, Li XO, Xie Y, Chen XP, Jiang JJ, Zha P, Hou JL, Gao ZL, Fan HM, Ding JG, Zhang DZ, Ren H. [HBsAg loss with Pegylated-interferon alfa-2a in hepatitis B patients with partial response to nucleos(t)-ide analog: new switch study]. Zhonghua Gan Zang Bing Za Zhi. 2018 Oct 20;26(10):756-764. doi: 10.3760/cma.j.issn.1007-3418.2018.10.005. Chinese. PMID 30481882
- [Derived] Hu P, Shang J, Zhang W, Gong G, Li Y, Chen X, Jiang J, Xie Q, Dou X, Sun Y, Li Y, Liu Y, Liu G, Mao D, Chi X, Tang H, Li X, Xie Y, Chen X, Jiang J, Zhao P, Hou J, Gao Z, Fan H, Ding J, Zhang D, Ren H. HBsAg Loss with Peg-interferon Alfa-2a in Hepatitis B Patients with Partial Response to Nucleos(t)ide Analog: New Switch Study. J Clin Transl Hepatol. 2018 Mar 28;6(1):25-34. doi: 10.14218/JCTH.2017.00072. Epub 2018 Mar 17. PMID 29577029